CLINICAL TRIAL: NCT06933563
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients With Relapsed / Refractory Myasthenia Gravis
Brief Title: UCAR T-cell Therapy Targeting CD19/BCMA in Patients With r/r Myasthenia Gravis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai Xiniao Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH-ZY-03
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Myasthenia Gravis
Keywords: Universal Allogeneic CAR T-cells; CD19/BCMA CAR T-cells
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-CD19/BCMA CAR T-cells (Experimental): Universal allogeneic CD19/BCMA CAR T-cells
  Interventions: Biological: UCAR T-cell group

INTERVENTIONS:
Biological: UCAR T-cell group — A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with relapsed or refractory Myasthenia gravis. This study aims to evaluate the safety and efficacy of the treatment with universal CD19/BCMA CAR T-cells.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal CD19/BCMA CAR T-cells in Relapsed or Refractory Myasthenia gravis.

Study intervention consists of a single infusion of universal CAR T-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when participants finish the visit 90 days after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Flow cytometry detected positive B cell CD19 or BCMA in the patient's peripheral blood.
3. Patients with relapsed refractory myasthenia gravis (MG) who have positive abnormal antibodies, the total score of MG-ADL ≥5, and the eye muscle score < 50% of the total score; It is classified as Grade II-IV according to the 2020 MGFA diagnostic criteria.
4. Specific requirements include: i. Receiving standardized treatment with at least one immunosuppressant for more than 1 year, and having any of the following malcontrolled conditions: 1) persistent inability to affect daily life; 2) Aggravation of MG symptoms and/or crisis episodes occur despite standard treatment; 3) Inability to tolerate immunosuppressive therapy. ii. plasma exchange or maintenance of intravenous immunoglobulin therapy is required.
5. Functional requirements for major organs are as follows:

   1. The bone marrow function needs to meet: a Neutrophil count ≥ 1.5× 10 ^ 9/L; b. Hemoglobin ≥90g/L: c. Platelets ≥ 80 × 10 ^ 9/L.
   2. Liver function: ALT ≤ 3 × UL; AST ≤ 3×ULN# Total bilirubin ≤ 2.0 ×ULN (excluding Gilbert syndrome, total bilirubin ≤ 3.0 × ULN).
   3. Renal function: creatinine clearance rate (CrCl) ≥ 30 ml/min(Cockcroft/Gault formula, excluding acute CrCl decline caused by the disease itself).
6. Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
7. Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Subjects with a history of severe drug allergies or allergic tendencies.
2. Presence or suspicion of uncontrolled or treatment-required fungal,bacterial, viral, or other infections.
3. Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis).
4. Subjects with insufficient cardiac function.
5. Subjects with congenital immunoglobulin deficiencies.
6. History of malignancy within five years.
7. Subjects with end-stage renal failure.
8. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer higher than the upper limit of detection; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing.
9. Subjects with psychiatric disorders and severe cognitive impairments.
10. Subjects who had participated in other clinical trials within 3 months prior to enrollment.
11. Subjects who have used immunosuppressive agents or biologics with therapeutic effects on the disease within five half-life before enrollment
12. Pregnant women or women planning to conceive
13. Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After UCAR T-cell Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 90 days After UCAR T-cell Infusion
Changes of Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | Up to 24 Months After UCAR T-cell Infusion
  MG-ADL scale assesses the impact of gMG on daily functions by measuring 8 signs or symptoms that are commonly affected in MG. Each item is measured on a 4-point scale, where a score of 0 represents normal function and a score of 3 represents the loss of ability to perform that function. Total scores range from 0 to 24 points, with a higher score showing more severe MG.
Quantitative Myasthenia Gravis Score (QMG) | Up to 24 Months After UCAR T-cell Infusion
  The QMG score is a 13-item scale used to quantify disease severity in myasthenia gravis. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No